CLINICAL TRIAL: NCT02032758
Title: Golfer's Cramp: Correlation of Wrist Movements and Surface EMG With Putter Movements
Brief Title: Study of Arm and Putter Movement in Golfers With Golfer's Cramp
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Charles Adler, Professor of Neurolgy, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 12-007930
Record Dates: First submitted 2014-01-02; First posted 2014-01-10 (Estimated); Results first posted 2016-07-25 (Estimated); Last update posted 2016-07-25 (Estimated); Status verified 2016-06

CONDITIONS: Occupational; Cramp(s)
Keywords: Occupational; Cramp(s)
MeSH Terms: conditions — Dystonic Disorders | interventions — Propranolol; Electromyography

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Golfers With Golfer's Cramp (Experimental): Subjects in this arm will be tested with the Opal device, the Science and Motion PuttLab (SAM), and the Surface Electromyography (EMG) to collect movement parameters while putting before and after a single dose of 10 mg Propranolol.
  Interventions: Drug: Propranolol; Device: Opal Device; Procedure: Science and Motion PuttLab (SAM); Device: Surface Electromyography EMG
- Golf Pros (Other): Subjects in this arm will be tested with the Opal device, the Science and Motion PuttLab (SAM), and the Surface Electromyography (EMG) to collect movement parameters while putting. The subjects in this arm will not receive any study drug.
  Interventions: Device: Opal Device; Procedure: Science and Motion PuttLab (SAM); Device: Surface Electromyography EMG

INTERVENTIONS:
Drug: Propranolol — Single oral dose of 10 mg propranolol
  Other Names: Inderal
  Arms: Golfers With Golfer's Cramp
Device: Opal Device — The Opal Device (APDM, Inc.) will be used to measure wrist movement.
Procedure: Science and Motion PuttLab (SAM) — The SAM will be used to study putter stroke movement and ball movement.
Device: Surface Electromyography EMG — The surface EMG will be used to evaluate co-contraction of the wrist flexor/extensor muscle groups and the wrist pronator/supinator muscle groups.

SUMMARY:
The investigators will investigate golfers with visual evidence of an involuntary movement while putting before and after treatment with a low dose of propranolol.

DETAILED DESCRIPTION:
Dystonia affecting athletes has received little research attention and there has been a lack of awareness or interest among both physicians and athletes. Task-specific dystonias or occupational cramps affect people while writing, typing, and or playing a musical instrument. Our group has previously shown that a subset of golfers who complain of the yips appear to have a task-specific dystonia or golfer's cramp. The yips are characterized by an inability to appropriately complete a golf stroke, most often putting and chipping strokes. Most individuals with the yips describe a jerking or shaking movement that interrupts their swing. In many cases the yips are disabling and the golfer, including professional tour players, give up golfing.

Golfers who have evidence of golfer's cramp will putt a series of putts during which they will be monitored for arm movements and putter movements. They will then be treated with a low dose of propranolol to see if there is a change in these parameters.

ELIGIBILITY:
Inclusion criteria:

* Age 18-75
* Complaint of golfer's cramp/yips
* Visual evidence of a movement disorder during putting
* Able to complete 80 putts during the session

Exclusion criteria:

* Contraindication to treatment with propranolol
* Movement disorder not when putting

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2014-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Charles Adler, MD, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Arizona, Scottsdale, Arizona, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from Mayo Clinic in Arizona.
Period: Overall Study
Arm/Group | Golfers With Golfer's Cramp | Golf Pros
Started | 27 | 11
Completed | 27 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Golfers With Golfer's Cramp | Golf Pros | Total
Number analyzed (Participants) | 27 | 11 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 11 | 27
  >=65 years | 11 | 0 | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 25 | 6 | 31
Region of Enrollment [Number; unit: participants]
  United States | 27 | 11 | 38

OUTCOME MEASURES:

1. Primary Outcome: Mean Dynamic Change of Rotation at Impact
Description: "Dynamic change of rotation at impact" is the velocity of rotation of the putter from the start of the forward swing until the time of impact with the golf ball.
Time Frame: baseline, approximately 45 minutes after propranolol dosing
Population: This variable was measured at baseline and then again approximately 45 minutes after propranolol in the group with golfer's cramp on the same day. The pro golfers did not take propranolol so they were only tested once, at baseline.
Measure: Mean (Standard Deviation); unit: degrees/sec
Arm/Group | Golfers With Golfer's Cramp | Golf Pros
Number analyzed (Participants) | 27 | 11
degrees/sec
  No propranolol | -38.4 (26.1) | -32.5 (9.8)
  After propranolol | -36.5 (36.5) | NA (NA) — The pro golfers did not take propranolol so they were only tested once, at baseline.

2. Secondary Outcome: Mean Total Putter Face Rotation Before Impact
Description: "Total putter face rotation before impact" is the degrees of rotation of the putter from the start of the forward swing until the time of impact with the golf ball.
Time Frame: baseline, approximately 45 minutes after propranolol dosing
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Golfers With Golfer's Cramp | Golf Pros
Number analyzed (Participants) | 27 | 11
degrees
  No propranolol | 3.3 (1.3) | 3.1 (0.6)
  After propranolol | 3.4 (1.9) | NA (NA) — The pro golfers did not take propranolol so they were only tested once, at baseline.

ADVERSE EVENTS:
Time Frame: Participants were monitored for adverse events on the day of the study.
Arm/Group | Golfers With Golfer's Cramp | Golf Pros
Serious Adverse Events (participants affected / at risk) | 0/27 | 0/11
Other Adverse Events (participants affected / at risk) | 0/27 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes